CLINICAL TRIAL: NCT03254030
Title: Does Careful Inspection of Colonic Mucosa During Insertion and Withdrawal During Bowel Scope Improve Rate of Adenoma Detection?
Brief Title: Does Inspection of Colonic Mucosa During Insertion Improve Adenoma Detection?
Acronym: INWARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD16/117
Record Dates: First submitted 2017-08-17; First posted 2017-08-18 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Adenoma Colon; Serrated Adenoma
Keywords: Adenoma; Sessile serrated adenoma
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Intervention Model Description: Participants are randomised to undergo the flexible sigmoidoscopy screening examination either for control or intervention group. Control group is to undergo inspection of colonic mucosa only during withdrawal phase of the examination. Intervention group will undergo the examination during which the colonic mucosa will be inspected during inspection and withdrawal phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspection on withdrawal (Placebo Comparator): Participants colonic mucosa will be examined only during withdrawal phase of the examination.
  Interventions: Other: Colonic inspection
- Inspection on insertion and withdrawal (Active Comparator): Participants colonic mucosa will be examined during insertion and withdrawal phase of the examination
  Interventions: Other: Colonic inspection

INTERVENTIONS:
Other: Colonic inspection — Participants who are randomised to undergo the intervention will have the colonic mucosa examined during inspection and withdrawal phase of examination
  Other Names: Inspection of colonic mucosa during insertion and withdrawal

SUMMARY:
This is a prospective randomised controlled trial to assess an intervention of inspection during both phases of colonoscopic examination ( insertion and withdrawal) improve adenoma detection rate when compared to inspection only during withdrawal.

DETAILED DESCRIPTION:
Successful implementation of colorectal screening programmes and improvement in colonoscopic technology have resulted in significant decrease in colorectal cancer incidence and mortality. Effectiveness of colonoscopy largely depends on detection and removal of adenomas before they become cancerous. Despite the vast improvement in colonoscopy training and technology, it remains as an imperfect tool. It has been reported that the adenoma miss rate during colonoscopy varies between 6-27% in clinical practice. Adenoma Detection Rate (ADR) is a surrogate marker of efficient colonoscopy. Researchers continue to explore various methods and technologies to improve adenoma detection such as frequent position changes, routine use of antispasmodics and devices to improve the mucosal visibility (third eye retro view scope, Transparent cap, Endocuff).

However, all the techniques are focused on the withdrawal stage of the examination. Colonic examination is traditionally performed with rapid passage of colonoscope to the caecum and a careful examination of mucosa is carried out during the withdrawal phase. Polyps are removed during the withdrawal phase. It is well known from expert opinion that some polyps are detected during the insertion phase rather than withdrawal phase especially in sigmoid and transverse colon. This could be due to different anatomical configuration of colon during insertion and withdrawal.

During insertion phase colonic mucosa is stretched and the folds are splayed due to the formation of loops and angulation hence affects the visualised area of the mucosa ahead of the colonoscope. During withdrawal, the colon is shortened and the adjacent folds are brought closer to each other. On withdrawal colon is much straighter. Therefore, it may expose different portions of colonic mucosal surface on insertion and withdrawal.

Flexible sigmoidoscopy Bowel cancer screening programme (Bowel Scope) has been successfully implemented since May 2013. Initial reports suggest ADR within Bowel Scope screening varies considerably.

Therefore, we propose a simple technique to improve ADR in Bowel Scope Screening.

RATIONALE FOR CURRENT STUDY

Recent report suggests that ADR within Bowel Scope screening (BSS) varies considerably. We propose a small technical alteration to improve ADR in BSS. A recent prospective trial highlighted that if polypectomy was performed only during Withdrawal Phase (WP) when compared to performing careful inspection and polypectomy during Inspection Phase (IP) plus WP, polyps could be missed in about 7% of patients. We hypothesised that careful inspection and polypectomy during both phases would be complementary and it would increase ADR by complete visualisation of recto sigmoid mucosa during Bowel Scope.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are referred for a bowel scope screening procedure

Exclusion Criteria:

* Patients lacking capacity to give informed consent
* Pregnant women
* Age less than 55 years
* Uncorrectable coagulopathy
* Patients who are not fit for flexible sigmoidoscopy
* Incomplete procedure

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 8 months
  Number of participants with at least one adenoma

SECONDARY OUTCOMES:
Polyp detection rate | 8 months
  Number of patients with at least one polyp
Mean number of adenoma per patient | 8 months
  Number of adenomas divided by the number of patients in that group
Total procedure time | 8 months
  Time taken to complete the procedure
Advanced adenoma detection rate | 8 months
  Number of patients with adenoma larger than 10mm and or consists of villous histology or high grade dysplasia

CONTACTS AND LOCATIONS:
Overall Officials: Rajaratnam Rameshshanker, MBBS,MRCP, Principal Investigator — London North West Healthcare NHS Trust
Locations (1):
- NorthWest London Hospitals - NOrthwick park hospital, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No